CLINICAL TRIAL: NCT01992731
Title: IUI vs. IVF/ICSI in Women Aged 38-42 Years: a Prospective Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Michael De Brucker, MD, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUI versus IVF/ICSI
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Infertility
Keywords: Age (38-42 years); pregnancy rates; 3 IUI cycles; 1 IVF/ICSI cycle
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IUI group (Active Comparator): Group 1: Patients undergo a standard treatment with 3 consecutive gonadotrophin stimulated IUI cycles Intervention: treatment choice and drug:(Follitropine Bèta, Puregon, MSD).
  vs.
  Interventions: Other: Drug: Follitropine Bèta
- IVF/ICSI arm (Active Comparator): Group 2: 1 Patients start immediately with IVF/ICSI instead of IUI. A standard antagonist protocol with treatment with a recombinant FSH (Follitropine Bèta, Puregon, MSD) is used.
  Intervention: treatment choice and drug: recombinant FSH (Follitropine Bèta, Puregon,
  Interventions: Other: Drug: Follitropine Bèta

INTERVENTIONS:
Other: Drug: Follitropine Bèta

SUMMARY:
Prospective randomised controlled trial: 3 IUI cycles versus 1 IVF/ICSI cycle in women aged 38-42 years.

DETAILED DESCRIPTION:
Study design:

Prospective randomised controlled trial: 3 IUI cycles versus 1 IVF/ICSI cycle in women aged 38-42 years. .

Group 1: 3 consecutive gonadotrophin stimulated IUI cycles (Follitropine Bèta, Puregon, MSD).

vs. Group 2: 1 IVF/ ICSI cycle - Recombinant FSH (Follitropine Bèta, Puregon, MSD) - Antagonist protocol.

ELIGIBILITY:
Inclusion Criteria:

Women aged between 38 and 42 years. Sperm: use of donor sperm or husband sperm reaching WHO criteria 2010.

Exclusion Criteria:

* Tubal infertility (even one tube).
* Major uterine or ovarian abnormalities
* Metabolic abnormalities

Ages: 38 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks
  Study design:
  Prospective randomised controlled trial: 3 IUI cycles versus 1 IVF/ICSI cycle in women aged 38-42 years.
  Group 1: 3 consecutive gonadotrophin stimulated IUI cycles (Follitropine Bèta, Puregon, MSD).
  vs. Group 2: 1 IVF/ ICSI cycle - Recombinant FSH (Follitropine Bèta, Puregon, MSD) - Antagonist protocol.
  Primary endpoint:
  Comparison of the cumulative ongoing pregnancy rates after 3 IUI cycles versus 1 IVF/ICSI cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Michael De Brucker, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UniversitairZB, Jette, Belgium